CLINICAL TRIAL: NCT01671631
Title: The Diastolic Pressure Gradient for Patients With Acute Coronary Syndrome: Evaluation of Non Culprit Lesions
Acronym: FORECAST
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Magna Graecia (Other)
Responsible Party: Principal Investigator, Ciro Indolfi, Professor, University Magna Graecia
Other Study IDs: FORECAST
Record Dates: First submitted 2012-08-20; First posted 2012-08-23 (Estimated); Last update posted 2012-08-23 (Estimated); Status verified 2012-08

CONDITIONS: Functional Evaluation of Non Culprit Lesions in ACS Patients

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Acute Coronary Syndrome: Patients with Acute Coronary Syndrome and multivessel coronary artery disease undergoing functional evaluation of non-culprit lesions.
  Interventions: Other: Measurement of intracoronary pressure

INTERVENTIONS:
Other: Measurement of intracoronary pressure

SUMMARY:
The assessment of non-culprit stenoses is an important issue in ACS. Adenosine administration is currently required for functional evaluation of stenosis severity using the fractional flow reserve (FFR). An alternative adenosine-independent index of coronary stenosis, the instantaneous wave-free ratio (iFR), was recently introduced.

Aim of the present study will be to evaluate the trans-stenotic instantaneous wave-free pressure gradient (iFG), the instantaneous wave-free ratio (iFR) and the fractional flow reserve (FFR) in ACS patients.

ELIGIBILITY:
Inclusion Criteria:

* age 40 to 80 years
* recent Acute Coronary Syndrome
* indication for coronary angiography
* presence of at least one non-culprit lesion requiring functional evaluation with fractional flow reserve (FFR):

Exclusion Criteria:

* Haemodynamically significant valvular disease
* controindication for Adenosin administration
* previous CABG on the index vessel

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with Acute Coronary Syndrome and multivessel coronary artery disease.
Sampling Method: Probability Sample

CONTACTS AND LOCATIONS:
Locations (1):
- Cardiologia Interventistica UMG, Catanzaro, Calabria, Italy

REFERENCES:
- See also: Web site, Division of Cardiology at Magna graecia University — http://www.cardiologia.unicz.it
- See also: Web site, Dipartimento di Scienze Mediche e Chirurgiche, Magna Graecia University — http://www.dsmc.unicz.it